CLINICAL TRIAL: NCT06256536
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase Ib/IIa Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of GZR18 Injection in Chinese Obese/Overweight Patients
Brief Title: A Study of GZR18 Injection in Chinese Obese/Overweight Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gan and Lee Pharmaceuticals, USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GL-GLP-CH2002
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GZR18 (Experimental): GZR18 injection s.c.
  Interventions: Drug: GZR18
- Placebo (Placebo Comparator): Placebo injection s.c.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GZR18 — 0.6 mg-30 mg
  Arms: GZR18
Other: Placebo — administered the same volume as GZR18
  Arms: Placebo

SUMMARY:
The study was a multicenter, randomized, double-blind, placebo-controlled phase Ib/IIa clinical study to evaluate the safety, tolerability, pharmacokinetics and efficacy of GZR18 injection in Chinese adult obese/overweight patients. This study is divided into Part A and Part B, which are to be conducted simultaneously.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female aged 18-65 years (inclusive);

  2. Obese subjects: BMI ≥ 28.0 kg/m2; or overweight subjects: 24.0 ≤ BMI < 28.0 kg/m2 with at least one comorbidity;

  3. Able to understand the procedures and methods in this study; willing to complete the study in strict accordance with the clinical study protocol and sign the ICF voluntarily.

Exclusion Criteria:

* 1. Suspicion that the subject may be allergic to any study drug or ingredient or congener from the investigator.

  2. Subjects with body weight change > 5.0% for any reason (diet, exercise, etc.) within 12 weeks prior to screening.

  3. Heart rate < 50 beats/min or > 100 beats/min on 12-lead ECG at screening.

  4. Presence of the following clinically significant 12-lead ECG abnormalities at screening.

  5. Alcohol abuse within 6 months prior to screening, or reluctance to stop alcohol abuse throughout the study, or a positive breath alcohol test result at screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2023-10-22 (Actual); Study Completion 2023-10-22 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events and serious adverse events | 38 weeks
Changes in weight from baseline to the end of treatment | 35 weeks

SECONDARY OUTCOMES:
trough concentrations following consecutive doses | 35 weeks
Changes in Body mass index (BMI) from baseline to the end of treatment | 35 weeks
Changes in Percentage of reduction in weight (%) from baseline to the end of treatment | 35 weeks
Changes in Waist circumference from baseline to the end of treatment | 35 weeks
Proportion of subjects with ≥5% reduction in body weight from baseline. | 35 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Liyuan Zhao, Ph.D, Study Director — Gan & Lee Pharmaceuticals.
Locations (1):
- Gan & Lee Pharmaceuticals Co., Ltd, Beijing, China